CLINICAL TRIAL: NCT02355912
Title: Adaptive Recalibration of Prosthetic Leg Neural Control System
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shirley Ryan AbilityLab (Other)
Responsible Party: Principal Investigator, Levi Hargrove, Director, Neural Engineering for Prosthetics and Orthotics Laboratory, Shirley Ryan AbilityLab
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: STU00101767
Record Dates: First submitted 2015-01-16; First posted 2015-02-04 (Estimated); Last update posted 2020-10-28 (Actual); Status verified 2020-10

CONDITIONS: Amputation
Keywords: Transfemoral

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Evaluate a real-time adaptive neural control system (Experimental): The prosthesis will be tuned, for each subject: level-ground walking, walking up and down slopes and walking up and down stairs. We anticipate that participants will visit the laboratory approximately 6-9 times over 2 months (2-3 visits for socket duplications and modifications, 2-3 visits for control system tuning, and an additional 2-3 visits for practice using the tuned system). By the end of these visits, the goal is to have a properly fitting socket and for the subjects to ambulate proficiently with the powered prosthesis. After tuning, the subjects will complete 20 ambulation circuits (level ground walking, walking up and down slopes, up and down stairs). This will provide training data for our pattern recognition control systems.
  Interventions: Device: Powered knee and ankle prosthesis

INTERVENTIONS:
Device: Powered knee and ankle prosthesis — A powered knee and ankle prosthesis developed by Vanderbilt University.

SUMMARY:
The purpose of this study is for transfemoral amputees to walk with an experimental robotic prosthesis. Electric signals will be measured from their muscles and used to help control an artificial leg. The investigators will record from sensors placed on a prosthesis and electric signals measured from muscles in the participants leg to see if the investigators can develop better computer programs to help predict subject actions and prostheses function.

DETAILED DESCRIPTION:
The investigators propose to use a powered knee-ankle prosthesis that is not yet commercially available. The hierarchical control framework the investigators are developing will be equally applicable to any prosthetic leg that needs to be transitioned between ambulation modes, including microprocessor-controlled passive devices.

The overall objective is to develop and evaluate an adaptive framework for controlling lower limb prostheses that compensates for changes in EMG signals. When a participant walks on a lower limb prosthesis, the output of the high-level controller (or ambulation mode predictor) directly influences patterns generated by the participant. After the participant has completed the subsequent stride, a gait pattern estimator (GPE), will provide a label of what the participant actually did. This may differ from the ambulation mode predictor output if there was a misclassification. The label will then be used to update the ambulation mode predictor algorithm such that future steps are predicted with higher accuracies. Finally, the resulting system will be transferred to an embedded system and tested in real-time with transfemoral amputees and compared to a non-adaptive system.

ELIGIBILITY:
Amputee Subjects

Inclusion Criteria:

* Lower Limb Amputees
* K2/K3/K4 ambulators

Exclusion Criteria:

* Over 250lbs body weight
* Inactive, physically unfit
* cognitive deficits or visual impairment that would impair their ability to give informed consent or to follow simple instructions during the experiments
* Pregnant women
* co-morbidity that interferes with the study (e.g. stroke, pace maker placement, severe ischemia cardiac disease, etc.)

Able-bodied Subjects:

Inclusion Criteria:

* no injury on either lower extremity

Exclusion Criteria:

* inactive, physically unfit
* over 250 lbs body weight
* cognitive deficits or visual impairment that would impair their ability to give informed consent or impair their ability to follow simple instructions during the experiments
* Pregnant women (status determined by self-reporting)
* co-morbidity that interferes with the study (e.g. stroke, pace maker placement, severe ischemia cardiac disease, etc.)

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-01; Primary Completion 2020-01 (Actual); Study Completion 2020-01 (Actual)

PRIMARY OUTCOMES:
Decreased error rates for pattern recognition system used to predict ambulation modes | Assessed at approximately 2 months and 6 months after enrollment
  Pattern recognition algorithms have been used to allow seamless and automatic transitioning between ambulation modes. Classification errors result in the prosthesis predicting the wrong ambulation mode. A decrease in errors results in improved mode prediction by the prosthesis. EMG from the participant and mechanical sensor data from the prosthesis are processed with the use of a phase-based-dependent pattern recognition classification method. The data collection will yield three groups of 10 real-time trials. The investigators primary analysis will be a repeated measures ANOVA with a planned contrast between the groups. The investigators will also complete a secondary analysis using the data collected while the participants ambulated outside of the laboratory. The total number of misclassifications will be computed. This will allow the investigator to evaluate the rate at which the overall classification system adapted.

CONTACTS AND LOCATIONS:
Overall Officials: Levi Hargrove, PhD, Principal Investigator — Shirley Ryan AbilityLab
Locations (1):
- Rehabilitation Institute of Chicago, Chicago, Illinois, United States